CLINICAL TRIAL: NCT04199559
Title: Evaluating Combination Therapy Using Autologous Dendritic Cells Pulsed With Antigen Peptides and Nivolumab for Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Evaluating Combination Therapy Using Autologous Dendritic Cells Pulsed With Antigen Peptides and Nivolumab for Subjects With Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Cttq (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019111810
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: NSCLC
MeSH Terms: interventions — Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous dendritic cells pulsed with antigen (Experimental): peptide(WT1-H/K-HELP, Survivin-H/K-HELP,MAGE-A4-H ⁄ K-HELP and MUC1-22) . Each dose contains of 10 million activated autologous DCs. Route of Administration: Intradermal.
  Interventions: Drug: Autologous dendritic cells pulsed with antigen

INTERVENTIONS:
Drug: Autologous dendritic cells pulsed with antigen — peptide(WT1-H/K-HELP, Survivin-H/K-HELP,MAGE-A4-H ⁄ K-HELP and MUC1-22) . Each dose contains of 10 million activated autologous DCs. Route of Administration: Intradermal

SUMMARY:
Study Arms: Patients receive autologous dendritic cells pulsed with antigen peptides ID on days 15, 29, 43,57,71,99,127and 155, and nivolumab IV over 60 minutes on days 15, 29, 43,57,71,85 99 and 113.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors are increasingly drawing much attention in the therapeutic development for cancer treatment. However, many cancer patients do not respond to treatments with immune checkpoint inhibitors, partly because of the lack of tumor-infiltrating effector T cells. DC vaccine may prime patients for treatments with immune checkpoint inhibitors by inducing effector T-cell infiltration into the tumors and immune checkpoint signals. The combination of DC vaccine and an immune checkpoint inhibitor may function synergistically to induce more effective antitumor immune responses, and clinical trials to test the combination are currently needed.

ELIGIBILITY:
Inclusion Criteria:

1. Be 20 years of age or older on day of signing informed consent.
2. Non-small cell lung cancer (NSCLC) patient with progression on or after platinum-based chemotherapy.
3. Have measurable disease based on Response Evaluation in Solid Tumors (RECIST) 1.1.
4. Have a performance status of 0 - 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
5. Life expectancy of >6 months.
6. Females of childbearing potential should have a negative urine or serum pregnancy.
7. Serum glutamate pyruvate transaminase (SGPT) =< 4.0 times upper limits of normal (ULN)
8. Serum glutamic-oxaloacetic transaminase (SGOT) =< 4.0 times ULN
9. Creatinine =< 2 times ULN
10. Patients who have one of the following HLA types: A2402, A0201, A0206
11. Pre-Leukaphersis evaluation
12. Hemoglobin > 10 g/dL (100 g/L)
13. White blood cell count 3.0-11.0 x 10^3/mm^3 (3.0-11.0 x 10^9/L)
14. Absolute granulocyte count >= 1.5 x 10^3/mm^3 (1.5 x 10^9/L)
15. Absolute lymphocyte count >= 1.0 x 10^3/mm^3 (1.0 x 10^9/L)
16. Platelet count >= 100 x 10^3/mm^3 (100 x 10^9/L)

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid or any other form of immunosuppressive therapy.
3. Hypersensitivity to nivolumab or any of its excipients.
4. Has a known additional malignancy.
5. Any diagnosis of autoimmune disease.
6. Pregnant or breastfeeding within the projected duration of the trial, starting with screening visit through the last dose of trial treatment.
7. Positive HIV-1, -2, or HTLV-1, -2, tests.
8. Positive HBV or HCV tests.
9. Positive syphilis tests.
10. Recipient of organ allografts.
11. Inability or unwillingness to return for required visits and follow-up exams.
12. Acute infection: any active viral, bacterial, or fungal infection that requires specific therapy.
13. Active uncontrolled infection, such as a sexually transmitted disease (STD), herpes, uncontrolled tuberculosis, malaria, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause
Disease Control Rate (DCR) | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zibing Wang, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China